CLINICAL TRIAL: NCT01447134
Title: Phase II Study of [18F]RGD-K5 in Head and Neck Cancer Patients
Brief Title: RGD-K5 in Head and Neck Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzu-Chen Yen, Department of Nuclear Medicine, Chang Gung Memorial Hospital
Other Study IDs: IRB99-3338A
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Surgical: Group (a) [Those to undergo surgical excision or biopsy] patients will receive RGD-K5 scan within two weeks of conventional image evaluations. The image result will be confirmed with histopathological results.
- Chemotherapy concurrent Radiation: Group (b) patients [Those with N2c-3M0 disease to receive chemotherapy followed by concurrent chemoradiotherapy] will receive RGD-K5 scan prior to beginning of the therapy, after induction chemotherapy, within two weeks after concurrent chemoradiotherapy and two months after completion of concurrent chemoradiotherpy; all within two weeks of conventional image evaluations.
- RGD-K5 scan: Group (c) patients [Those with M1 disease to receive biotherapy or chemotherapy] will receive RGD-K5 scan prior to the beginning of the first line systemic therapy, two weeks after beginning of the first line systemic therapy, within two weeks of first response evaluation for the first line systemic therapy, and within two weeks after end of the first line systemic therapy; each RGD-K5 scan would be performed within two weeks of conventional image studies. The systemic therapy might be biotherapy or chemotherapy.

SUMMARY:
1. Primary endpoint(s): To determine the relationship between the drug distribution and angiogenesis in head and neck cancer patients.
2. Secondary endpoint(s): To expand the safety database of [F-18]RGD-K5 and to correlate the parameters from the image study to clinical treatment response and prognosis.

DETAILED DESCRIPTION:
This is an uncontrolled, open-labeled, non-randomized, prospective study. The study duration is expected to be completed in a period of 3 year. Up to 100 patients would be included. Group A would be those to undergo surgical excision or biopsy (n=20); Group B would be those with N2c-3M0 disease to receive chemotherapy followed by concurrent chemoradiotherapy (n=40); and Group C would be those with M1 disease to receive biotherapy or chemotherapy (n=40). Group A patients could be included into Group B or C if qualified. Each participant must fulfill all the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients (including nasopharyngeal cancer)
* Age equals or more than 20 years old
* Referred by Chang Gung Memorial Hospital (CGMH) Head and Neck Oncology team.
* Willing to sign the informed consent

Exclusion Criteria:

* Patient who is pregnant or lactating;
* Patients with a concomitant or previous 2nd primary cancer other than head and neck malignancy;
* Unable to tolerate MR or PET/CT scan, such as those with magnetic implants (e.g. those received intracranial aneurysm surgery, cardiac pacemaker, artificial valves replacement, artificial ears), poor blood sugar control (fasting sugar more than 200 mg/dl), claustrophobia, unable to lie still.
* Unable to give informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 patients would be included. Group A would be those to undergo surgical excision or biopsy (n=20); Group B would be those with N2c-3M0 disease to receive chemotherapy followed by concurrent chemoradiotherapy (n=40); and Group C would be those with M1 disease to receive biotherapy or chemotherapy (n=40). Group A patients could be included into Group B or C if qualified.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)